CLINICAL TRIAL: NCT01499992
Title: Rehabilitation of Reconstructed Shoulder Rotator Cuff : Optimizing Physical Therapy Dosage and Effect of Aquatic Physical Therapy - A Randomized, Factorial Study
Brief Title: Rehabilitation of Reconstructed Shoulder Rotator Cuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Joy MacDermid, Co-Director HULC Clinical Research lab, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18466
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2012-01

CONDITIONS: Full Thickness Rotator Cuff Tear
Keywords: Shoulder rehabilitation; Rotator cuff tear; Physiotherapy; aqua therapy; Therapy dosage; adjunctive aquatic physical therapy
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aquatic physical therapy (Experimental): aquatic physical therapy program which will be conducted twice weekly for 10 weeks and will include a 40-50 minute hydrotherapy session emphasizing range of motion and light resistive exercises of the arm, primarily focussing on the shoulder.
  Interventions: Procedure: Standard physical therapy program PLUS aquatic physical therapy; Other: standard care
- standard care (No Intervention)

INTERVENTIONS:
Procedure: Standard physical therapy program PLUS aquatic physical therapy — 2. Standard physical therapy program PLUS aquatic physical therapy: The above PLUS a aquatic physical therapy program which will be conducted twice weekly for 10 weeks and will include a 40-50 minute hydrotherapy session emphasizing range of motion and light resistive exercises of the arm, primarily focusing on the shoulder. The program will start with general mobility of the other upper limb joints to allow time for preconditioning of the painful shoulder. Shoulder exercises will emphasize flexion, rotation and abduction and a slow transition from pain-free range to the restricted range of motion to maximize the effectiveness of the heat and buoyancy.
  Arms: aquatic physical therapy
Other: standard care — Total of 12 weeks; each exercise session will be 20 -30 minutes of direct contact and additional supervised exercise as defined by assignment and stage.
  Arms: aquatic physical therapy

SUMMARY:
The aim of this study to define the optimal rehabilitation for clients with full thickness rotator cuff reconstruction, with two goals: 1. Finding the optimal physical therapy dosage in enhancing post-operative outcomes of shoulder pain, shoulder joint range of motion, shoulder muscle strength, upper extremity function; and 2. Finding the effect of aquatic physical therapy in enhancing the post-operative outcomes.

DETAILED DESCRIPTION:
Measurement devices:

Biodex: Biodex system is a muscle strength testing and rehabilitation instrument used in the testing and rehabilitation services for shoulder, elbow, wrist, hip, knee and ankle. Modes of operation for exercise and testing include isokinetic, passive, isometric, isotonic, and reactive eccentric. Patients are tested for their muscle performance for the required number of repetitions in the required mode. The muscle performance is measured by calculating the average peak torque (in Nm) and analyzed across the group of patients.

Goniometer: A manual devise used to measure joint range of motion. Visual Analogue Scale: A scale with 0 to 10, with 0 being no pain, and 10 being severe pain.

Measurement procedure:

All the subjects posted for surgery will be tested prior to and again 6 weeks following surgery for:

Shoulder Pain is measured using a visual analog scale. Shoulder Range of motion is measured using a standard goniometer. Shoulder Muscle performances are measured using Biodex.

ELIGIBILITY:
Inclusion Criteria:

* full thickness rotator cuff tear treated by arthroscopic or mini-open repair by a specialized upper extremity surgeons
* mentally competent
* able to read and write
* able to return for follow-up
* 18-65 years old

Exclusion Criteria:

* associated surgical procedures (Concomitant fractures, capsular releases surgical decompression)
* nerve injury
* neurological conditions
* irreparable massive rotator cuff tear, and
* comorbid health problems that limit rehabilitation potential (Rheumatoid arthritis, Diabetes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
strength | 3 month after the surgery

SECONDARY OUTCOMES:
patient satisfaction | 3 and 6 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joy MacDernmid, PhD, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- St Joseph's health Care London, London, Ontario, Canada

REFERENCES:
- [Background] Ellenbecker TS, Sueyoshi T, Winters M, Zeman D. Descriptive report of shoulder range of motion and rotational strength six and 12 weeks following arthroscopic superior labral repair. N Am J Sports Phys Ther. 2008 May;3(2):95-106. PMID 21509132
- [Result] Roddey TS, Olson SL, Gartsman GM, Hanten WP, Cook KF. A randomized controlled trial comparing 2 instructional approaches to home exercise instruction following arthroscopic full-thickness rotator cuff repair surgery. J Orthop Sports Phys Ther. 2002 Nov;32(11):548-59. doi: 10.2519/jospt.2002.32.11.548. PMID 12449254